CLINICAL TRIAL: NCT03063190
Title: Evaluation of Cholecalciferol Supplementation in Chronic Kidney Disease Patients With Restless Leg Syndrome
Brief Title: Cholecalciferol Supplementation in Restless Leg Syndrome in Patients With Chronic Kidney Disease
Acronym: RLS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: the main research is no longer in the Institution
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLS vitamin D
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2019-10

CONDITIONS: Restless Leg Disorder; Renal Disease Bone; Renal Disease, End Stage; Hyperparathyroidism, Secondary; Adynamic Bone Disease; Vitamin D Deficiency
MeSH Terms: conditions — Restless Legs Syndrome; Chronic Kidney Disease-Mineral and Bone Disorder; Kidney Failure, Chronic; Hyperparathyroidism, Secondary; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hyperparathyroidism_0 (Placebo Comparator): Chronic Kidney Disease patients with parathyroid hormone higher than 300pg/ml
  Interventions: Drug: Placebo Oral Tablet
- Hyperparathyroidism_1 (Active Comparator): Chronic Kidney Disease patients with parathyroid hormone higher than 300pg/ml
  Interventions: Drug: Vitamin D
- Adynamic_0 (Placebo Comparator): Chronic Kidney Disease patients with parathyroid hormone lower than 150pg/ml
  Interventions: Drug: Placebo Oral Tablet
- Adynamic_1 (Active Comparator): Chronic Kidney Disease patients with parathyroid hormone lower than 150pg/ml
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — patients will receive vitamin D supplementation according to guidelines
  Arms: Adynamic_1; Hyperparathyroidism_1
Drug: Placebo Oral Tablet — patients will receive placebo oral tablets
  Arms: Adynamic_0; Hyperparathyroidism_0

SUMMARY:
Restless leg syndrome (RLS) is sleep disorder characterized by an unpleasant feeling in the lower limbs, which can be accompanied by paresthesias, and need for urgent movement of the legs. Its diagnosis is clinical, based on an International Committee of the Study of RLS (International Restless Legs Syndrome Study) questionnaire. Its prevalence is about 5-15% in the general population, being twice as frequent in women and with a tendency to increase incidence with aging. In the chronic kidney disease (CKD) population, mainly in patients on dialysis, the prevalence increases by up to 70%. Vitamin D deficiency is associated with RLS and active vitamin D supplementation seems to improve RLS and severity. It is seems, studies on the role of vitamin D supplementation in CKD population are missing. The clinical-scientific hypothesis of this study is that replacement of vitamin D (cholecalciferol) will improve the symptoms of RLS. As parathyroidectomy can relieve RLS, the aim of researchers is to randomize patients with CKD on dialysis to receive cholecalciferol or placebo in 2 distinct groups: secondary hyperparathyroidism and adynamic bone disease.

ELIGIBILITY:
Inclusion Criteria

- adult patients with chronic kidney disease on dialysis, with vitamin D deficiency.

Exclusion Criteria

* current treatment for restless leg syndrome
* history of parathyroidectomy in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-31 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Improvement RLS severity | 6 months
  Reduction of the disease's symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No